CLINICAL TRIAL: NCT04946292
Title: Developing and Evaluating a Theory-derived Intervention to Improve Oral Health of Community-dwelling Elderly
Brief Title: Empowering Older Adults for Healthy Living and Better Dental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Gao Xiaoli, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R-221-000-140-133
Record Dates: First submitted 2021-06-07; First posted 2021-06-30 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Diseases; Dental Caries
Keywords: oral health; health behaviours; periodontal disease; theory-derived intervention
MeSH Terms: conditions — Periodontal Diseases; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory-derived intervention (Experimental): Questionnaire will be used including the scales for three dominant theoretical models, Health Belief Model (HBM), Theory of planned behaviour (TPB) and Social Cognitive Theory (SCT). The theoretical model that best explains the health behaviours of the selected participants will be selected for designing oral health intervention.The theory-derived intervention will address the constructs/domains of the selected model(s) in the context of the three target behaviours (diet, toothbrushing and dental flossing).
  Interventions: Behavioral: Theory-derived intervention
- Conventional health education (Active Comparator): Participants will be randomly assigned to the control group, stratified by gender and education level. Allocation concealment will be ensured by using sealed opaque envelopes.
  Interventions: Behavioral: Conventional health education

INTERVENTIONS:
Behavioral: Theory-derived intervention — The intervention will be delivered through multimedia materials and group activities, as appropriate. Participants will spend approximately 30-45 minutes for the intervention. Intervention materials and activities will be carefully designed to address all the constructs/ domains of the selected theoretical model(s). The effectiveness of the interventions will be evaluated using behavioural outcomes (diet, brushing, flossing) and clinical outcomes (oral hygiene, caries and periodontal conditions).
  Arms: Theory-derived intervention
Behavioral: Conventional health education — The conventional health education will be delivered through an oral health talk and oral health booklet. Topics covered are: (i) common oral diseases and its consequences; (ii) common dental problems among older adults; (iii) importance of oral health measures (healthy diet, toothbrushing and dental flossing); and (iv) proper techniques for toothbrushing and dental flossing.
  Arms: Conventional health education

SUMMARY:
Ageing of the world's population is accelerating. Despite the health challenges they face, older people should not be stereotyped as frail and dependent. Healthy ageing is possible if adequate care is provided and effective intervention is delivered for healthy living. Common oral diseases (dental caries and periodontal diseases) are determined to a great extent by health behaviours (diet and oral hygiene) and are controllable through effective interventions. Hence, this study aims to test the theoretical models for health promotion, develop theory-derived intervention, and evaluate its effectiveness in improving oral health of older adults. The study hypothesis is that theory-derived intervention is more effective than conventional health education in eliciting positive behaviours and controlling oral diseases in older adults.

DETAILED DESCRIPTION:
This study targets older adults and aims to (i) test the explanatory power of the dominant theoretical models/ frameworks, (ii) develop theory-derived intervention, and (iii) evaluate the effectiveness of the theory-derived intervention. The hypothesis is that theoretical-derived intervention is more effective than conventional health education in improving oral health behaviours and preventing oral diseases among older adults.

The sample size needed for this study was calculated by using the software G*Power version 3.1.9.2 (Franz Faul, University of Kiel, Germany). The sample size calculation was based on the primary outcomes, namely increment of coronal caries and increment of root caries, and independent t-tests for comparing means of two independent groups. A caries incidence study among the elderly reported that the mean (SD) 5-year caries incidence were 2.65 (3.14) for coronal caries and 2.21 (2.83) for root caries 17. The 2-year incidence of coronal caries and root caries were therefore estimated to be 1.06 (1.26) and 0.88 (1.13), respectively, in the control group. The effect of an intervention is considered clinically significant if it reduces the caries incidence by 40%. Based on a significance level of 5% and a power of 80%, 140 subjects per group are needed for coronal caries and 165 subjects are needed for root caries outcome measures. To take both outcome measures into account, the higher number (i.e., n=165) will be adopted. Allowing for a 25% attrition rate, 220 elderly persons will need to be recruited into each group, giving a total sample size of 440.

Each participant will be required to complete a detailed questionnaire at the initial visit through face-to-face interviews. Information on socio-demographic background (gender, age, education level, past occupation, and type of housing) and oral health behaviours (diet, toothbrushing and dental flossing) will be collected. The questionnaire will also include the scales for three dominant theoretical models, namely, Health Belief Model (HBM), Theory of planned behaviour (TPB) and Social Cognitive Theory (SCT).

The theoretical model that best explains the health behaviours will be selected for designing oral health intervention. Intervention materials and activities will be carefully designed to address all the constructs/ domains of the selected theoretical model(s). Relevant medical literatures will be referred to. The needs, interest, and health literary of the target group (i.e. older adults of varied social and educational backgrounds) will be taken into full consideration. The intervention will be tested in a small group of 15-20 older people to ensure its relevance, practicality, and acceptability.

Participants will be randomly assigned to two groups, stratified by gender and education level. Allocation concealment will be ensured by using sealed opaque envelopes. The two groups will receive conventional health education and theory-derived intervention, respectively.

At baseline and 6-, 12-, and 24-months post-intervention, each participant will a) undergo an oral examination (dental checkup) by a trained dentist, who will be calibrated against an experienced oral epidemiologist and blinded to the group allocation, and b) complete a questionnaire (detailed questionnaire at baseline and short questionnaire for follow-ups). Chi-square tests will be used for comparing proportions. Parametric or non-parametric methods will be adopted for comparing means. ANCOVA (analysis of covariance) and multiple regressions will be performed to evaluate the effects of various factors on the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 55-70 years old
* Living in the community (alone or with family members), instead of residing in a nursing home
* Having at least 8 natural teeth
* No plan to immigrate in 3 years

Exclusion Criteria:

• Life-threatening disease; impaired cognitive function (e.g. Alzheimer's syndrome); radiotherapy in the head and neck region

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Increment of coronal caries | From baseline to 2 years post-intervention
  Number of new surfaces with coronal caries
Increment of root caries | From baseline to 2 years post-intervention
  Number of new surfaces with root caries

SECONDARY OUTCOMES:
Change in dietary behaviours (favourable/unfavourable) | From baseline to 2 years post-intervention
  Using a questionnaire, dietary behaviours will be categorised into:
  1. favourable (frequency of snack intake, sweet/desert intake and/or sugary drinks <2times/day)
  2. unfavourable (frequency of snack intake, sweet/desert intake and/or sugary drinks >=2times/day)
Change in toothbrushing behaviours (favourable/unfavourable) | From baseline to 2 years post-intervention
  Using a questionnaire, toothbrushing behaviours will be categorised as:
  1. favourable (frequency of brushing >=2times/day)
  2. unfavourable (frequency of brushing <2times/day)
Change in flossing behaviours (favourable/unfavourable) | From baseline to 2 years post-intervention
  Using questionnaire to evaluate frequency of flossing (with >=once/day considered as favourable and <once/day considered unfavourable)
Change in oral hygiene status (plaque score) | From baseline to 2 years post-intervention
  Presence or absence of dental plaque on tooth surfaces
Change in periodontal condition | From baseline to 2 years post-intervention
  Number of sites with deep periodontal pockets, shallow periodontal pockets, and gingival bleeding only

CONTACTS AND LOCATIONS:
Overall Officials: Gao Xiaoli, PhD, Principal Investigator — Faculty of Dentistry, National University of Singapore
Locations (1):
- Faculty of Dentistry, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao X, Wong ML, Kalhan AC, Xie JJ, Siti Hajar H, Yeo ABK, Allen PF. Theory-derived intervention to improve oral health of older adults: study protocol for a randomised controlled trial. BMJ Open. 2022 Dec 12;12(12):e064791. doi: 10.1136/bmjopen-2022-064791. PMID 36523250